CLINICAL TRIAL: NCT07289152
Title: Pediatric Health Empowerment: Improving Children´s Perioperative Experiences With Patient-Reported Measures
Brief Title: Pediatric Anesthesia: The Childs Voice
Acronym: PHEASE
Status: Recruiting | Type: Observational
Sponsor: Gødstrup Hospital (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1-16-02-129-25
Record Dates: First submitted 2025-12-03; First posted 2025-12-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-05

CONDITIONS: Pediatric Anesthesia; Pediatric Surgery; PROMs; PREMs
Keywords: PROM; Patient-reported outcom measues; Children; child; PREM; Patient-reported experience measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children age 4-12, undergoing surgery and general anesthesia

SUMMARY:
In Denmark, around 25,000 children under 18 undergo general anesthesia annually. Hospital stays and anesthesia can induce significant anxiety and stress in children due to unfamiliar environments, procedures, and communication issues. This anxiety can be linked to postoperative complications such as emergence delirium and may negatively impact both the child and their family's well-being. Engaging patients actively in their healthcare, including pediatric cases, is essential for improving outcomes. Assessing perioperative patient and family outcomes, particularly through patient-reported outcome measures (PROM) and patient-reported experience measures (PREM), can significantly enhance the quality of care provided to children. While PROMs are widely used in adults, they are less common in pediatric settings. The Pediatric Scale for Quality of Recovery (PedSQoR), developed by Australian and American researchers, is one such tool designed to measure recovery in children. This study aims to translate andvalidate the PedSQoR for Danish children aged 4-12. Furthermore, no existing instruments comprehensively assess pediatric surgery patients' experiences under general anesthesia, particularly from the child's perspective without relying on parents as proxies. Empowering children to express their healthcare experiences gives healthcare workers an insight into what matters for children and gives children a more positive outlook on healthcare, benefiting lifelong engagement.

Study Aims and Objectives: The study aims to enhance the assessment of children's outcomes and experiences in perioperative settings, ultimately improving pediatric perioperative healthcare. The objectives include:

1. Translation and Adaptation: a. Translate and adapt the PedSQoR for Danish children aged 4-12. b. Validate the Danish PedSQoR version.
2. Development of a PREM Instrument: a. Develop a comprehensive PREM for children's experiences during surgery and anesthesia. b. Pilot-test and adjust the PREM questionnaire with a group of children aged 4-12.

Study Methods:

1. PedSQoR Translation and Validation:

   A single-center prospective cohort study will adapt and test the PedSQoR for Danish children. The process involves translating the 21-item scale, validating it with a sample size of 150, and ensuring reliability through various statistical methods, including Cronbach's Alpha and test-retest reliability. Data will be collected from the Department of Anesthesiology and Intensive Care at Gødstrup Hospital.
2. PREM Instrument Development:

This study will develop a PREM instrument using the Warwick Patient Experiences Framework (WaPEF), which encompasses seven dimensions of patient experience. The process will involve forming a panel of child experts, conducting focus groups, and translating insights into a pictorial questionnaire. The PREM will undergo pilot testing with 20 children to validate its effectiveness in capturing the dimensions of the WaPEF.

Research Ethics: Given the vulnerability of children in research, this study will prioritize their safety and comfort, ensuring the study's benefits outweigh any potential risks. Informed consent will be obtained from both parents and children. The study will be registered with the Region Central Denmark's list of research projects and will not require approval from the Scientific Ethics Committee.

DETAILED DESCRIPTION:
Project title: Pediatric Healthcare Empowerment: Improving Children's Perioperative Experiences with Patient-Reported Measures Acronym: PHEASE

Impact:

Understanding and improving children's experiences is integral to enhancing pediatric healthcare services. Annually, approximately 6 million children worldwide undergo general anesthesia, and the potential impact on their well-being and behavior is significant. The hospital environment, inadequate communication with staff and negative postoperative experiences can contribute to anxiety and sadness, particularly due to a lack of insight into children's unique needs. The common practice of relaying information to parents or caretakers often results in the child's perspective being overlooked. This study promises to empower 4-12-year-olds to express their thoughts to enhance the perioperative experience. This study will translate a newly developed tool for measuring patient-reported outcome measures in Pediatric Scale for Quality of Recovery (PedSQoR) and create a tool for children to express their experiences so that hospital staff can improve the quality of care. The impact extends beyond immediate outcomes, with the potential for lifelong benefits for children shaping their healthcare experiences. Background In Denmark, 25,000 children under the age of 18 undergo general anesthesia annually (1).

Admission to hospitals and general anaesthesia affect children; a hospital stay can cause a child to experience anxiety about procedures, unknown environments, pain and fasting (2).

Poor communication with staff may negatively influence the mood and behavior of the child (3). Furthermore, postoperative anxiety and melancholy may be linked to the onset of emergence delirium, the disconcerting hospital setting, and a limited understanding of the unique requirements of children (4). Post-operative symptoms can impose a burden on both children and their parents, potentially requiring them to take sick leave for varying durations. However actively engaging patients in their healthcare experience improves health outcomes, a principle applicable to pediatric cases as well (5). Consequently, assessing perioperative patient and family outcomes, postoperative well-being, and experiences may improve outcomes for children undergoing anesthesia. Ferreira et al. (2023) advocate for the combined use of patient-reported outcome measures (PROM) and patient-reported experience measures (PREM). This integrated approach incorporates both the objective and subjective aspects of the patient's experience. By 2 utilizing both measures in tandem, healthcare providers can gain a more nuanced and comprehensive insight into the overall quality of care from the patient's perspective (6).

PROMs are used widely in the adult population. Patient outcomes after surgery and anaesthesia can be assessed with the 15-item Quality of Recovery Score (QoR-15) (5). For children, a group of Australian researchers have developed a 21 item Pediatric Scale for Quality of Recovery (PedSQoR) measuring children´s recovery, this will be translated and validated into Danish (7). PREMs are tools that capture patients' perspectives on their interactions with healthcare services, including their experiences with the hospital environment and staff. Heath et al.

(2023) illustrate that children's experiences during a hospital stay can differ significantly from those of their parents. Therefore, children must have a direct and independent voice in the assessment of their care (2). Following the United Nations Convention on the Rights of the Child, every child is entitled to express their views on any matters affecting them. Ensuring their right to share insights regarding their experiences, particularly in the context of a hospital visit, it is crucial to enable children to provide input on their healthcare encounters, utilizing tools such as PROM and PREM (8). No instruments have been developed to validly assess patient experiences for pediatric surgery patients undergoing general anesthesia in children, and very few instruments exist to measure children's experiences without using parents as a proxy (3, 4, 6). Previous research has shown that empowering 4-12-year-olds to express their thoughts on enhancing and making the Operating Room less daunting for them has lifelong benefits (9). When children have a say in their healthcare experiences, they tend to develop a more positive outlook, leading to reduced fear and anxiety during medical visits, ultimately contributing to improved lifelong healthcare engagement (2, 10, 11). Aim The overall aim of this study is to enable the assessment of children's outcomes and experiences in the perioperative setting, ultimately contributing to improving all pediatric healthcare. Objectives

1. a. To translate and adapt the PedSQoR for Danish children aged 4-12.

1. b. To validate the Danish version of the PedSQoR in children aged 4-12.
2. a. To develop a comprehensive PREM for children's experiences during surgery and general anaesthesia.

2. b. To pilot-test and adjust the questionnaire on a group of children aged 4-12 who have undergone surgery and anaesthesia. 3 Methods Study 1 - Translating and adaptation of the PedSQoR for Danish children Study design: Adaption and clinimetric testing in a single-centered prospective cohort study.

Construction: Translated the PedSQoR for children into Danish, the 21 items will be validated. The rating scale will use a Likert scale and tested on 10 Danish children, to confirm the ranking (7). Inclusion criteria: Pediatric patients aged 4-12, American Society of Anesthesiologists physical status classification (ASA) I-III undergoing surgery in Gødstrup Hospital (12). Exclusion criteria: Children with cognitive or sensory disorders, children or parents who do not speak Danish, and patients for whom there is no consent to participate.

Setting: Department of Anesthesiology and Intensive Care at Gødstrup Hospital where we provide anaesthesia for 1050 children annually for a variety of surgical procedures within orthopaedics, urology, and general surgery. Data collection: Baseline data will be collected from the electronic medical journal and entered into Research Electronic Data Capture (REDCap) hosted at Aarhus University. The PedSQoR survey will be distributed by mail and entered into REDCap. Statistical method: Based on previous studies a sample size of 150 participants is needed to obtain reliable power (participation proportion 50%). Clinimetric validity will be tested by convergent, construct, and discriminant validity. Reliability will be tested with internal consistency based on Cronbach´s Alpha, and test and retest reliability will be analyzed.

Responsiveness will be assessed with the Cohen size effect and standardized response mean.

The completion rate will evaluate acceptability and feasibility and the mean times to complete the PedSQoR Danish. For analyzing data, we will use STATA version 17.0 BE.

Study 2. Development of a PREM instrument for children Study design: Development of a comprehensive measuring instrument for children's experiences during surgery and general anesthesia by using the Warwick Patient Experiences Framework (WaPEF) 7 dimensions, which includes Patients as active participants, Responsiveness of services, an Individualized approach, Lived experience, Continuity of care and relationships, Communication, Information, and Support. Development of items: The process will be guided by a panel of children recruited by the local Department of Pediatrics among their chronic patients. The panel will be considered experts having considerable experience with hospitals. We will conduct four focus group sessions involving a sample of 4-5 children of the same age who have undergone general anesthesia, and supplement data with individual interviews with children as needed. The interview guide will be developed to engage children in the conversation (13). All interviews will be recorded and transcribed. 4 Questionnaire Design: Based on insights from the interviews important themes and phrases will be translated into questions and answers on a pictorial questionnaire, incorporating the identified dimensions. Pilot testing and validation: Face validity of the questionnaire will be tested on 2-3 children through either in-person or telephone interviews and adjustments will be made if deemed necessary. After the adjustments, the questionnaire will be pilot tested on a group of 20 children, to validate if the questionnaire captures the children´s experiences according to the 7 dimensions of the WaPEF. The questionnaire will be administered on paper and data will be entered into REDCap. Inclusion criteria/ exclusion criteria/ setting: same as study 1. Data analysis: Transcripts from focus group interviews will be analysed using thematic analysis aligned with the 7 generic dimensions of WaPEF (14). Through collaborative efforts, the team will formulate consistent codes, subsequently applying them to the remaining two focus group transcripts using deductive coding. A comprehensive discussion within the research team will ascertain if the seven dimensions adequately encompass all emerging themes, resolving any discrepancies. Iterative modifications to the coding process will be made to ensure thorough coverage and prevent the oversight of any dimensions.

Expected papers

1. Translation and adaption of the PedSQoR for Danish children aged 4-12
2. Childrens experiences of surgery and anaesthesia. A focus group study
3. Development of a Pediatric Patient-Reported Experience Measurement Instrument for children aged 4-12 undergoing anesthesia and surgery Research ethics Given their vulnerability in research, children necessitate careful consideration to ensure the study neither harms nor burdens them, weighing this against the study's significance in empowering children's voices. Therefore, specialized communication strategies will be employed in interactions with children. All interviews will be carried out by the PhD student who is a highly experienced nurse anesthetist with long experience in communication with children. Informed written consent will be sought from both parents and children. The study does not mandate approval from the Scientific Ethics Committee but will be registered on the Region Central Denmark's list of research projects.

5

Organization of the project The project will be conducted at Gødstrup Hospital, with Anne Højager Nielsen Ph.D., MCN, Associate Professor serving as the main supervisor.

Co-supervisors: Veronica Pisinger Ph.D. and researcher at the National Institute of Public Health; Denmark has special insight into the validation of questionnaires. Associate Professor and nurse anesthetist Pether Jildenståhl from Lunds University, Sweden has special insight into anaesthesia and children's needs and rights.

Collaborators: A/Prof Paul Lee-Archer, BMedSci, MBBS, FANZCA, MMed(ClinEpi), PhD, Senior Staff Specialist, Anaesthesia, Queensland Children's Hospital, Associate Professor, Faculty of Medicine, University of Queensland, and Professor Andrew Davidson FAHMS, Medical Director, Melbourne Childrens Trail Centre, Murdoch Children Research Institute,will host the international research stay.

Pediatric anesthetists and staff at Gødstrup Hospital. The PhD student: Draft of the protocol, data collection, data management, and data analysis.

The manuscripts will be drafted by the Ph.D. student, who will be the primary author of all publications. The PhD student will present research findings at conferences and international events. The PhD student will disseminate Relevant results to patient organizations and the public.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 4-12, American Society of
* Anesthesiologists physical status classification (ASA) I-III
* undergoing surgery

Exclusion Criteria:

* Children with cognitive or sensory disorders
* children or parents who do not speak Danish,
* patients for whom there is no consent to participate.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children undergoing surgery and general anesthesia aged 4-12 years.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
To validate the Danish version of the PedSQoR in children aged 4-12. | From enrollment to the end of week 4 after surgery
To pilot-test and adjust the questionnaire on a group of children aged 4-12 who have undergone surgery and anaesthesia | From enrollment to 4 weeks after surgery
  Patient Reported Experience Measure (PREM)

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (4):
  - Aarhus University Hospital, Aarhus, Central Jutland
  - Aalborg University Hospital, Aalborg, Region North
  - Copenhagen University Hospital, Copenhagen, Region Sjælland
  - Gødstrup Hospital, Herning

IPD SHARING:
Plan to Share IPD: Undecided